CLINICAL TRIAL: NCT02130037
Title: The Effect Size of Cognitive Behavioral Therapy Via a Smartphone Application on Bulimia Nervosa and Binge Eating Disorder Symptoms
Brief Title: Cognitive Behavioral Therapy Via a Smartphone Application on Bulimia Nervosa and Binge Eating Disorder Symptoms
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no grants
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Eitan Gur MD, MD, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-14-1001-EG-CTIL
Record Dates: First submitted 2014-05-01; First posted 2014-05-02 (Estimated); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: B.E.D AND BULIMIA PATIENT; SMARTPHONE OWNER; BASIC ENGLISH SPEAKER
Keywords: APPLICATION; SMARTPHONE; BULIMIA; B.E.D; BINGE EATING DISORDER
MeSH Terms: conditions — Bulimia; Binge-Eating Disorder | interventions — Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- psychotherapy only (Active Comparator)
  Interventions: Other: psychotherapy
- application (Experimental)
  Interventions: Behavioral: application; Other: psychotherapy

INTERVENTIONS:
Behavioral: application — along standard psychotharpy we use a smartphone application that allows the patient to monitor her meals, behaviours, emotions and thoughts and to communicate them directly in real time to their therapists.
  Other Names: recovery record
  Arms: application
Other: psychotherapy — standard psychotherapy for eating disorders

SUMMARY:
Background: research show that cognitive behavioral therapy (CBT) is effective inreducing bulimia nervosa (BN) and binge eating disorder's (BED) symptoms. Today, with the development of technology there are efforts being made for developinga treatment to these eating disorders threw the media, most of these attempts are based on the CBT method. The size of the effect that CBT given threw the internet has on BN and BED is still not entirely clear. Research presented today are mostly based on treatments that were given threw email or Skypeor an automatic self- help stage program. These researches show heterogenic results about the effect it had on eating disorders. In this research we aim to investigate the effect size that a CBT treatment threw a smartphone application that combines a clinician online reply and an automatic feedback in addition to astandard ones a week clinic treatment has on BN and BED symptoms frequency.

Methods: Our aim is to make a research using an application that treats that offers an automatic and human therapist and dietitian reply threw a similar application that is suited for them. A selected 40 BN or sub-threshold BN or BED patients, men and women ages 18-60 ,that will turn to the "Sheba eating disorder medical center" will include the research. Half of the participants will receive aCBT treatment threw a smartphone application along with astandardclinical treatment that includes ones a week session with a therapist and ones a week session with a dietitian and the other half will receive a standardclinic treatment alone. We will test the eating disorder symptoms using eating disorders questionnaires at the starting point, at the end of a six months treatment and six months after finishing the treatment.

Importance: This research will allow testing the need and benefit that a personal and direct patient- therapist connection has over a standardones a week meeting connection format. In addition, treating with a web application in the future might have a benefit of saving time spent on getting to the clinic, will allow to shorten the time of the session in the clinic and will save cost of the face to face treatment.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of binge eating disorder
* clinical diagnosis of bulimia
* smrtphone owner
* english speaker

Exclusion Criteria:

* clinical diagnosis of type 1 diabetes
* clinical diagnosis of other axis 1 psychological problems
* pregnancy
* clinical diagnosis of celiac disease

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2015-06 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
EDI-2 REDUCED SCORE | BEFORE INTERVANTION, AFTER INTERVANTION, 6 MONTHES AFTER INTERVANTION

SECONDARY OUTCOMES:
EAT-26 REDUCED SCORES | BEFORE INTERVANTION, AFTER INTERVANTION, 6 MONTHES AFTER INTERVANTION

CONTACTS AND LOCATIONS:
Overall Officials: EITAN GUR, MD, Principal Investigator — Director of the Eating Disorder Dept.Sheba Medical Center Tel Hashomer; NIR BEN YOHANA, MA, Study Director — Eating Disorder Dept. Sheba Medical Center Tel Hashomer; SHIR ZILBERSHTAIN, BA, Study Chair — Eating Disorder Dept.Sheba Medical Center Tel Hashomer; MICHAL WOHL-LOTAN, PHD, Study Chair — Eating Disorder Dept. Sheba Medical Center Tel Hashomer
Locations (1):
- Eating Disorder Dept.Sheba Medical Center Tel Hashomer, Ramat Gan, Tel Hashomer, Israel